CLINICAL TRIAL: NCT06883773
Title: Does Engagement in a Computerized M-Health Intervention Increase With Digital Rewards?
Brief Title: Digital Rewards and Retention in a M-health App
Acronym: DIGITALRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Cezar Giosan, Associate Professor of Psychology, University of Bucharest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DIGITALGAMINGRCT
Record Dates: First submitted 2025-02-24; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Transdiagnostic Psychopathology; Attrition; Engagement; Depression, Anxiety; Stress
Keywords: crypto; digital rewards; mHealth; attrition; CBT; NFT
MeSH Terms: conditions — Tooth Wear; Depression; Anxiety Disorders; Cryptococcosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crypto reward group (Experimental): The participants will be enrolled in a weekly, 6 module intervention, which will require them to read psychoeducational materials, complete quizzes regarding those materials, complete the module-specific exercise, and then get rewarded in cryptocurrency. The participants will be assessed before, during and after the intervention.
  Interventions: Behavioral: Multipurpose Online Tool
- Sweepstakes reward group (Active Comparator): The participants will be enrolled in a weekly, 6 module intervention, which will require them to read psychoeducational materials, complete quizzes regarding those materials, complete the module-specific exercise, and then earn the chance to win vouchers for an online store. The participants will be assessed before, during and after the intervention.
  Interventions: Behavioral: Multipurpose Online Tool
- Waitlist (Other): The participants will be enrolled on the platform, but only for completing the assessments.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Multipurpose Online Tool — The intervention consists of 6 psychoeducational modules, on the Canvas teaching platform. They are automated, requiring no interaction with others (except for communication between participants and the team). Participants go through the psychoeducational modules, then do the corresponding exercise, and then access their rewards (if they belong to the experimental or comparative groups).
  Arms: Crypto reward group; Sweepstakes reward group
Other: No intervention — The participants will be assessed but without any intervention
  Arms: Waitlist

SUMMARY:
Attrition and user engagement are two challenges that eHealth interventions struggle with. Attempts to address this have been previously made through gamification, instructional design and using different types of incentives. Overall, any type of reward, be it non-financial or monetary is better than the controls, but the latter usually produce a greater effect. It is also worth mentioning that having an affective value attached to the reward itself is also important to user retention and engagement. Given the ever-increasing interest in cryptocurrency and its current relevance, the present study - a randomized clinical trial with three arms - aims to compare cryptocurrency to non-monetary rewards regarding their effectiveness in reducing attrition and increasing engagement. In order to do this, a mental-health computerized intervention will be developed, in which the users will have to complete several modules, during which time they will be rewarded either with cryptocurrency, sweepstake rewards (e.g., vouchers), or nothing.

DETAILED DESCRIPTION:
Albeit effective, eHealth interventions suffer from very high dropout rates. Finding novel ways in which to maximise user retention and engagement in such settings can be beneficial, and exploring cryptocurrency as a potential reward may be worthwhile, since motivation seems to increase as the reward is perceived as more meaningful by the recipient.

The design is experimental, between-subjects, with one independent variable (the type of reward offered) and mental health (e.g., depression, anxiety, stress, and transdiagnostic constructs) as well as engagement and retention outcomes. Thus, three groups will be formed: two in which participants will be enrolled in the modular MOTO intervention and will receive different rewards, and one in which they will not receive any intervention or reward but will be evaluated as part of a waitlist control group. The modular MOTO intervention involves, in addition to the mentioned assessments, the completion of six weekly modules, each focused on specific aspects of mental health and containing exercises that may improve psychological well-being. These modules are automated, requiring no interaction with others (except for communication between participants and research team). Each of these modules contains the following: psychoeducational section(s) that participants must complete; a short test of 5-10 questions after each section to assess understanding of the material; (only for the first two groups); a link where they can obtain their rewards; the exercise corresponding to that module; the evaluation corresponding to that module.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Participant retention | From enrollment to the end of the 6 week intervention
  The numbers of participants that get to finish the entire intervention

SECONDARY OUTCOMES:
User Engagement Scale - Short Version (UES-SF) | From the first module to the last (from week 1 to 6)
  Score on how engaged the users feel while participating in the intervention - how satisfied and how much they value each intervention module.
  Minimum value = 1 Maximum value = 5 A higher score means a better outcome (i.e., a higher user engagement).
The Depression, Anxiety and Stress Scale (DASS-21) - Depression | On week 1 and week 6 of the intervention
  The users will be assessed to see if the intervention decreases depression symptoms.
  Minimum value = 0 Maximum value = 21 (raw score); please note that scores are usually doubled in order to maintain consistency with the DASS-42, which would result in a maximum of 42.
  Higher scores on this subscale are associated with a worse outcome (i.e. depression symptoms), and a total score can be compounded across all 3 subscales, after doubling their raw scores. This total score is a general psychological distress score.
The Depression, Anxiety and Stress Scale (DASS-21) - Anxiety | On week 1 and week 6 of the intervention
  The users will be assessed to see if the intervention decreases anxiety symptoms.
  Minimum value = 0 Maximum value = 21(raw score); please note that scores are usually doubled in order to maintain consistency with the DASS-42, which would result in a maximum of 42.
  Higher scores on this subscale are associated with a worse outcome (i.e. anxiety symptoms), and a total score can be compounded across all 3 subscales, after doubling their raw scores. This total score is a general psychological distress score.
The Depression, Anxiety and Stress Scale (DASS-21) - Stress | On week 1 and week 6 of the intervention
  The users will be assessed to see if the intervention decreases stress symptoms.
  Minimum value = 0 Maximum value = 21 (raw score); please note that scores are usually doubled in order to maintain consistency with the DASS-42, which would result in a maximum of 42.
  Higher scores on this subscale are associated with a worse outcome (i.e. stress symptoms), and a total score can be compounded across all 3 subscales, after doubling their raw scores. This total score is a general psychological distress score.
DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure-Adult | On week 1 and week 6 of the intervention
  This is a DSM-5-TR screener for symptoms, to provide additional information beyond the other secondary measures.
  Minimum score = 0 Maximum score = 8 (depression, mania, somatic symptoms, psychosis, repetitive thoughts and behaviors, personality functioning); 4 (anger, suicidal ideation, sleep problems, memory, dissociation); 12 (anxiety, substance use).
  A rating of mild (i.e., 2) or greater on any item within a domain (except for substance use, suicidal ideation, and psychosis) may serve as a guide for additional inquiry and follow up to determine if a more detailed assessment for that domain is necessary. For substance use, suicidal ideation, and psychosis, a rating of slight (i.e., 1) or greater on any item within the domain may serve as a guide for additional inquiry and follow-up to determine if a more detailed assessment is needed. A greater score is associated with a worse outcome.
The Intolerance of Uncertainty Scale: Short Version (IUS-12) | On week 1 and week 6 of the intervention
  This is a transdiagnostic mental health factor that describes an individual's distress and ability to negatively perceive uncertainty as a whole.
  Minimum score = 12 Maximum score = 60 A greater score is associated with a worse outcome (i.e., more intense intolerance of uncertainty)
The Difficulties in Emotion Regulation Scale: Brief Version (DERS-16) | On week 1 and week 6 of the intervention
  This is a transdiagnostic factor that describes a person's management and control of emotional states.
  Minimum score = 16 Maximum score = 80 A greater score is associated with a worse outcome (i.e., more difficulty in reglating emotions)
Ruminative Response Scale (RRS-10) | On week 1 and week 6 of the intervention
  This is a transdiagnostic factor that describes a person's tendency to continually focus on negative emotions, experiences and thoughts.
  Minimum score = 10 Maximum score = 40 A higher score is associated with a worse outcome (i.e., more intense ruminations)
Automatic Thoughts Questionnaire (Short Version) - ATQ -8 | On week 1 and week 6 of the intervention
  This is a transdiagnostic contruct that describes thoughts that occur spontaneously, triggered either by external or internal states of events.
  Minimum score = 8 Maximum score = 40 A higher score is associated with a worse outcome (i.e., greater frequency of negative automatic thoughts)
The Cognitive Fusion Questionnaire (CFQ-7) | On week 1 and week 6 of the intervention
  This is a transdiagnostic construct that measures how much people get entangled and immersed in their thoughts and beliefs.
  Minimum score = 7 Maximum score = 49 A higher score is associated with a worse outcome (i.e., a stronger tendency towards cognitive fusion, becoming more entangled with one's own internal experiences and thoughts)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bucharest, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided